CLINICAL TRIAL: NCT06061172
Title: Evaluation of a Digital Tool Enhancing GPs' Information Management in the Treatment of Patients with Multimorbidity - a Pilot Study (gp-multitool)
Brief Title: Digital Tool Enhancing GPs' Information Management for Patients with Multimorbidity - a Pilot Study
Acronym: gp-multitool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-100786-BO-ff
Record Dates: First submitted 2023-09-08; First posted 2023-09-29 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2023-12

CONDITIONS: Asthma; Breast Neoplasms; Coronary Disease; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Pulmonary Disease, Chronic Obstructive; Comorbidities and Coexisting Conditions
MeSH Terms: conditions — Asthma; Breast Neoplasms; Coronary Disease; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Participants are assigned to intervention group and control group, respectively, in parallel for the duration of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): Care as usual
- Intervention group (Experimental): GPs in the intervention arm have to use the web application for every patient at least twice (i.e., at least once a quarter), and have to use at least four specific questionnaires at least once, i.e. 1a is required, and either 2a or 2b, and either 3a or 3b, and either 4a or 4b or 4c. Results from the questionnaires need to be discussed between GPs and patients. Additionally, at least one medication review is obligatory.
  Interventions: Other: gp-multitool.de

INTERVENTIONS:
Other: gp-multitool.de — The intervention is based on a digital tool, which implements recommendations of the S3 guideline "multimorbidity" of the German College of General Practitioners and Family Physicians. The tool includes nine questionnaires addressing four dimensions of care:
  1. preferences (including a. treatment goals, and b. involvement of other persons in decision making);
  2. activities (including a. activities and participation, and b. social support);
  3. treatment (including a. problems with medication, and b. treatment burden);
  4. complaints (including a. pain, b. psychiatric disorders, and c. other complaints).
  The GPs can send the questionnaires by email to the patients and the patients can fill out the questionnaires at their home or in the waiting room of the GP's practice using their own smartphones, tablets or computers. The digital tool also includes instructions for conducting a medication review. Results from talks between GPs and patients can be documented in the tool.
  Arms: Intervention group

SUMMARY:
The gp-multitool.de study is a cluster-randomized controlled trial that aims to enhance evidence-based and patient-centered care for patients with multimorbidity by assessing and providing information relevant for the primary care of this patient group. This pilot study examines the feasibility of the gp-multitool.de study, i.e., intervention and evaluation in GP practices in urban and rural administrative districts in Germany.

DETAILED DESCRIPTION:
The gp-multitool.de study is a cluster-randomized controlled trial that enhances evidence-based and patient-centered care for patients with multimorbidity by assessing and providing information relevant for the primary care of this patient group. It aims to reduce the time patients spend in hospital (primary outcome) and their outpatient health care use, and to improve process quality of care, patients' health-related quality of life, and patient satisfaction (secondary outcomes).

This cluster-randomized controlled pilot study examines the feasibility of the gp-multitool.de study, i.e., intervention and evaluation in GP practices. Specifically, the aims of the pilot study are 1. to pilot the gp-multitool.de intervention over six months and to test acceptance, functionality, reliability and usability in general practices under real world conditions, 2. to assess feasibility of the study design, i.e., recruitment of practices and patients, baseline data acquisition, randomization, implementation of the intervention, and outcome data acquisition, and 3. to provide data for the final sample size calculation of the evaluation study.

GPs in the intervention group receive access to the digital tool, together with a brief introduction to its functionalities, a written manual, and contact data of a telephone support hotline, which can be called in case of any technical or organizational problems in relation to the digital tool. GPs in the control group receive no intervention and provide care as usual.

Patients will be recruited from GP practices in urban and rural administrative districts in Germany. The gp-multitool.de study is based on telephone interviews of patients and their GPs. Practices will be randomized after the baseline assessment by an independent statistician who does not have access to the assessed patient and practice data. The primary outcome will be analyzed using a multilevel mixed-effects negative-binomial regression model, and secondary outcomes will be analyzed by multilevel mixed-effects linear and negative-binomial regression models.

In addition to quantitative data collection, a qualitative process evaluation with all participating GPs and one patient from each practice will be conducted based on a pre-defined semi-structured interview guide. The process evaluation will focus on compliance with the study protocol, problems with functionality, usability and reliability of the tool and possible sources of bias in the study. The interviews will be digitally recorded, transcribed verbatim and analyzed by qualitative content analysis.

ELIGIBILITY:
Inclusion Criteria:

* participation in a DMP; in Germany, DMPs have been implemented in outpatient care for asthma, breast neoplasms, coronary heart disease, diabetes mellitus type 1, diabetes mellitus type 2, and chronic obstructive pulmonary disease
* at least two of the following coexisting conditions: Hypertension, Lipid metabolism disorders, Chronic low back pain, Severe vision reduction, Joint arthrosis, Diabetes mellitus, Chronic ischemic heart disease, Thyroid dysfunction, Cardiac arrhythmias, Obesity, Hyperuricemia/Gout, Prostatic hyperplasia, Lower limb varicosis, Liver diseases, Depression, Asthma/COPD, Gynaecological problems, Atherosclerosis/PAOD, Osteoporosis, Renal insufficiency, Cerebral ischemia/Chronic stroke, Cardiac insufficiency, Severe hearing loss, Chronic cholecystitis/Gallstones, Somatoform disorders, Hemorrhoids, Intestinal diverticulosis, Rheumatoid arthritis/Chronic polyarthritis, Cardiac valve disorders, Neuropathies, Dizziness, Dementias, Urinary incontinence, Urinary tract calculi, Anemias, Anxiety, Psoriasis, Migraine/chronic headache, Parkinson's disease, Cancers, Allergies, Chronic gastritis/GERD, Sexual dysfunction, Insomnia, Tobacco abuse, Hypotension

Exclusion Criteria:

* no capacity to consent
* functional limitations precluding participation in the intervention (eg, loss of vision)
* functional limitations precluding participation in telephone interviews (eg, loss of hearing)
* limited German language skills precluding participation in telephone interviews
* no access to a personal device with access to the internet (i.e., smartphone, tablet or personal computer)
* participation in other trials during the observation time of the pilot study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 123 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-08-29 (Actual)

PRIMARY OUTCOMES:
Time spent in hospital during the preceding six months | Once at baseline (before randomization of practices) and once at follow-up (immediately after the intervention)
  The outcome will be assessed by asking the patients how often they had been in hospital during the preceding six months and how many days each hospital stay lasted. The total time in hospital will be calculated by adding the duration of all stays together.

SECONDARY OUTCOMES:
The number of contacts with the GP during the preceding six months | Once at baseline (before randomization of practices) and once at follow-up (immediately after the intervention)
  The outcome will be assessed by asking the patients how often they had used their GP during the preceding six months.
The number of contacts with outpatient specialists during the preceding six months | Once at baseline (before randomization of practices) and once at follow-up (immediately after the intervention)
  The outcome will be assessed by asking the patients how often they had used outpatient specialists during the preceding six months.
The number of contacts with home care services during the preceding six months | Once at baseline (before randomization of practices) and once at follow-up (immediately after the intervention)
  The outcome will be assessed by asking the patients how often they had used home care services during the preceding six months.
Process quality of care as assessed by the summary score of the "GP-reported core set of quality indicators for older adults with multimorbidity in primary care" during the preceding six months | Once at baseline (before randomization of practices) and once at follow-up (immediately after the intervention)
  The outcome will be assessed by the "GP-reported core set of quality indicators for older adults with multimorbidity in primary care" (Schäfer I et al. 2023, DOI: https://doi.org/10.1186/s12916-023-02856-0), which has a possible range between 0 and 12 points. Higher scores indicate a better quality of primary care.
Process quality of care as assessed by the summary score of the "patient-reported core set of quality indicators for older adults with multimorbidity in primary care" during the preceding six months | Once at baseline (before randomization of practices) and once at follow-up (immediately after the intervention)
  The outcome will be assessed by the "Patient-reported core set of quality indicators for older adults with multimorbidity in primary care" (Schäfer I et al. 2023, DOI: https://doi.org/10.1186/s12916-023-02856-0), which has a possible range between 0 and 7 points. Higher scores indicate a better quality of primary care.
Self-rated health as assessed by the EuroQoL visual analogue scale | Once at baseline (before randomization of practices) and once at follow-up (immediately after the intervention)
  The outcome will be assessed by the EuroQoL visual analogue scale (Herdman M et al. 2011, DOI: 10.1007/s11136-011-9903-x), which has a possible range between 0 and 100 points. Higher scores indicate a better self-rated health.
Health-related quality of life as assessed by the "EuroQoL five dimension five level scale" descriptive system, German value set | Once at baseline (before randomization of practices) and once at follow-up (immediately after the intervention)
  The outcome will be assessed by the "EuroQoL five dimension five level scale" (EQ-5D-5L) descriptive system (Herdman M et al. 2011, DOI: 10.1007/s11136-011-9903-x). A summary score will be calculated using the German value set (Ludwig K et al. 2018, DOI: 10.1007/s40273-018-0615-8). According to the German value set, the EQ-5D descriptive system has a possible range between 1.0 and -0.661 points. Higher scores indicate a better health-related quality of life.
Patient satisfaction with organization of care as assessed by the European Task Force on Patient Evaluation of General Practice Care questionnaire | Once at baseline (before randomization of practices) and once at follow-up (immediately after the intervention)
  The outcome will be assessed by subscale 'organization of care' of the European Task Force on Patient Evaluation of General Practice Care questionnaire (EUROPEP, Wensing M et al. 2000, DOI: https://doi.org/10.3109/13814780009069953). The score has a possible range between 0 and 4 points each and higher values indicate higher patient satisfaction.
Patient satisfaction with clinical performance as assessed by the European Task Force on Patient Evaluation of General Practice Care questionnaire | Once at baseline (before randomization of practices) and once at follow-up (immediately after the intervention)
  The outcome will be assessed by subscale 'clinical performance' of the European Task Force on Patient Evaluation of General Practice Care questionnaire (EUROPEP, Wensing M et al. 2000, DOI: https://doi.org/10.3109/13814780009069953). The score has a possible range between 0 and 4 points each and higher values indicate higher patient satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ingmar Schäfer, PD Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data are available from the principal investigator upon reasonable request.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available from July 2025 until April 2027.
Access Criteria: Reasonable request, non-profit organisations.

REFERENCES:
- [Derived] Nothacker J, Paucke V, Lezius S, Zapf A, Luhmann D, Scherer M, Schafer I. Implementation of the German Clinical Practice Guideline for Multimorbidity Using a Digital Tool in Primary Care: Pilot Cluster Randomized Clinical Trial. JMIR Aging. 2025 Nov 20;8:e79767. doi: 10.2196/79767. PMID 41263476